CLINICAL TRIAL: NCT00533858
Title: Effect of Lacidipine and Losartan on 24 Hour Systolic Blood Pressure Variability in Elderly Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-2007-083
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension
Keywords: Systolic hypertension
MeSH Terms: conditions — Hypertension; Isolated Systolic Hypertension | interventions — lacidipine; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lacidipine (4 mg) or losartan (50 mg) — lacidipine (4 mg) or losartan (50 mg), both given once daily at the same hour in the morning (approximately at 8 AM) for 12 weeks

SUMMARY:
The aim of this study is to evaluate the effect of lacidipine and losartan in elderly hypertensive patients on reducing the 24 hour systolic BP variability, which is one of the potential parameter to consider in treating elderly hypertensive patients.

DETAILED DESCRIPTION:
In this study, we investigate the effects of two anti-hypertensive medications on systolic BP variability profile as a pilot study. This is a prospective, randomized, open-label, blinded end point (PROBE), parallel group study with two treatment arms. At the end of an initial 2-week washout period, during which any eventual anti-hypertensive drug is discontinued, patients fulfilling the inclusion criteria are randomly treated with the lacidipine (4 mg) or losartan (50 mg), both given once daily at the same hour in the morning (approximately at 8 AM) for 12 weeks. If the BP goal (SBP < 140 mmHg and DBP < 90 mmHg) has not been attained after 4 week's treatment, 12.5 mg hydrochlorothiazide (HCTS) once daily can be added.

Patients are checked 24-h ambulatory BP monitoring (ABPM) at the end of the washout period and after 12 weeks of active treatment. At each visit, seated cuff SBP and DBP, heart rate, use of concomitant medication and spontaneously reported adverse events are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age > 65 years)
* Essential hypertension (systolic BP > 140 mmHg or diastolic BP > 90 mm Hg)
* Provide written informed content

Exclusion Criteria:

* Secondary hypertension
* Myocardial infarction or cerebrovascular accident within the preceding 6 months
* Clinically significant valvular heart disease, heart failure (Class III, IV), renal insufficiency (serum creatinine > 2.5mg/dl), hepatic failure, uncontrolled diabetes mellitus
* Known hypersensitivity to the drugs used in the study.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-09; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
The change of 24-hour, one day systolic BP standard deviation (SD) within subjects (the difference of SD before and after 12 weeks' treatment) in lacidipine group and losartan group

SECONDARY OUTCOMES:
The change of 24-hour, one day diastolic BP standard deviation (SD) within subjects (the difference of SD before and after 12 weeks' treatment) in lacidipine group and losartan group
The difference of the changes in office diastolic and systolic BP after 12 weeks' treatment between lacidipine group and losartan group
The difference of the mean 24-hour ABPM systolic and diastolic BP after 12 weeks' treatment between lacidipine group and losartan group
The difference of the diastolic and systolic BP control rates after treatment between the 2 groups
The difference of the changes in 24-hour, one day BP standard deviation (SD) within subjects between lacidipine group and losartan group
The difference of the variation of coefficient (CV) of the mean values (24-hour BP SD divided by the mean multiplied by 100) between 2 groups
The difference of the smoothness index (SI, dividing the average of the 24 hourly change after treatment by the corresponding standard deviation) between 2 groups
The difference of the changes in pulse pressure after treatment between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Cheol-Ho Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Kyeonggi, South Korea